CLINICAL TRIAL: NCT00788944
Title: An Open-Label Study To Evaluate The Prevalence Of Phenotypic Poor Metabolizers At CYP2D6 Among Venlafaxine-Treated Outpatients With Depression
Brief Title: Determine The Percentage Of Depressed Outpatients Who Do Not Effectively Metabolize Extended-release Venlafaxine HCl
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0600B1-4433; B2411001
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Procedure: blood draw

INTERVENTIONS:
Procedure: blood draw — Test Article was not provided to subjects for this study.

SUMMARY:
This is a study to determine the percentage of patients with depression who are treated with extended-release venlafaxine HCl (U.S. marketed brand Effexor XR®) who are Poor Metabolizers (based on the levels of the drug in the blood) at 2D6 (a system in the liver that breaks down some medications and other chemicals).

ELIGIBILITY:
Inclusion Criteria:

* Men and women subjects aged 18 years or older.
* Current outpatient treatment with extended-release venlafaxine HCl (U.S. marketed brand Effexor XR®), within the US Food and Drug Administration (FDA)-approved dosage range for depression (37.5 mg/day to 225 mg/day), for 8 weeks or less.
* Ability to have a blood draw within 4 to 12 hours of the most recent dose of Effexor XR®.

Exclusion Criteria:

* Determination by the investigator that a blood draw is contraindicated.
* Participation in an investigational study within the past 30 days where the study medication is not known.
* Previous treatment with Effexor XR® or extended-release venlafaxine HCl (generic) in the 6 months prior to current treatment regimen.
* Treatment with DVS SR within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 971 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
0-desmethyl venlafaxine/venlafaxine ratio (levels of the drug in the blood) | 1 day

SECONDARY OUTCOMES:
Determine the percentage of patients treated with extended-release venlafaxine HCl who are genotypic Poor Metabolizers. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (49):
- United States (49):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Tuscon, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Temecula, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Cromwell, Connecticut
  - Pfizer Investigational Site, Milford, Connecticut
  - Pfizer Investigational Site, Coral Gables, Florida
  - Pfizer Investigational Site, Lauderhill, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Naperville, Illinois
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Florence, Kentucky
  - Pfizer Investigational Site, Columbia, Maryland
  - Pfizer Investigational Site, Pittsfield, Massachusetts
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Stevensville, Michigan
  - Pfizer Investigational Site, Chesterfield, Missouri
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, Kalispell, Montana
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Wilmington, North Carolina
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Mason, Ohio
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Bridgeville, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pottstown, Pennsylvania
  - Pfizer Investigational Site, Reading, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Bellevue, Washington

REFERENCES:
- [Derived] Preskorn SH, Kane CP, Lobello K, Nichols AI, Fayyad R, Buckley G, Focht K, Guico-Pabia CJ. Cytochrome P450 2D6 phenoconversion is common in patients being treated for depression: implications for personalized medicine. J Clin Psychiatry. 2013 Jun;74(6):614-21. doi: 10.4088/JCP.12m07807. Epub 2013 Mar 13. PMID 23541126
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0600B1-4433&StudyName=Determine%20The%20Percentage%20Of%20Depressed%20Outpatients%20Who%20Do%20Not%20Effectively%20Metabolize%20Extended-release%20Venlafaxine%20HCl